CLINICAL TRIAL: NCT06807697
Title: A Pilot Investigation of the Quality of Life Before and After Radiotherapy in Patients With Head and Neck Cancer
Brief Title: Quality of Life Before and After Radiotherapy in Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Jacopo Lanzetti, Doctor in Dental Hygiene, University of Turin, Italy
Other Study IDs: 00424
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Cancer; Quality of Life (QOL)
Keywords: Quality of Life; Head and Neck Cancer; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HNC and waiting to undergo curative radiotherapy
  Interventions: Radiation: Curative radiotherapy for Head and Neck Cancers

INTERVENTIONS:
Radiation: Curative radiotherapy for Head and Neck Cancers — Radiotherapy is a localized, non-invasive, painless therapy, mostly performed on an outpatient basis, capable of causing necrosis or the death of tumor cells through the use of high-energy radiation called ionizing radiation.

SUMMARY:
Worldwide, head and neck cancers (HNCs) are widespread (650,000 cases per year) and cause more than 330,000 deaths per year. Almost all cases, about 90%, are cancers of the oral cavity, oropharynx, and larynx.

In conventional clinical practice, HNCs are treated primarily with radiation therapy (RT), often used in combination with surgery and/or chemotherapy. Like most anti-neoplastic therapies, RT carries significant adverse effects both acute and chronic. Both types of adverse effects have a significant impact on quality of life (QoL).

The aim of the study is to examine the worsening of QoL in patients with HNC before and after cancer therapy and to assess the extent that each factor has in its worsening.

ELIGIBILITY:
Inclusion Criteria:

* patients between the ages of 18 and 75 years;
* patients who presented at their first dental visit with a diagnosis of HNC.

Exclusion Criteria:

* patients who had already undergone cancer therapies (excisional surgery or chemotherapy or radiation therapy) at the time of the first dental visit;
* patients with depression or social anxiety;
* patients with language difficulties.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Head and Neck Cancer and waiting to undergo curative radiotherapy. HNC patients attach great importance to their health-related quality of life. In addition, there is evidence that the QoL of HNC survivors is poorer than that of the general population due to the significant functional limitations caused by the disease and treatment, this is because the head and neck district is the site of several organs that play an important role in the basic functions of daily life, including breathing, speeching, chewing, and swallowing, and are important for appearance. Moreover, HNC leads to a high incidence of psychosocial problems among survivors, such as depression, social isolation, and addiction and substance abuse, which in turn post to negative consequences with regard to QoL.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
University of Washington Quality of Life Questionnaire version 4.1 | 1 month
  The UW-QOL v4.1 is a widely recognized questionnaire for reporting physical and socio-emotional dysfunction after HNC treatment and consists of short multifactorial questions specific to HNC and to assess the patient's perception of general QoL in the past 7 days. The questionnaire includes 12 questions to assess pain, appearance, activity, leisure, swallowing, chewing, speech, shoulder, taste, salivation, mood, and anxiety. There are two subdomains: physical and social-emotional. The physical function items are chewing, speech, swallowing, taste, saliva and appearance. Social function includes anxiety, mood, pain, activity, recreation, and shoulder function.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza, Torino, Italy

IPD SHARING:
Plan to Share IPD: Undecided